CLINICAL TRIAL: NCT05382806
Title: Reversal of Remimazolam by a Single Dose of Flumazenil After Monitored Anesthesia Care in Gynecological Ambulatory Surgery: a Prospective Randomized Controlled Trial
Brief Title: Reversal of Remimazolam by a Single Dose of Flumazenil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Yea-Ji Lee, Professor, Konkuk University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KUMC2021-11-058
Record Dates: First submitted 2022-05-11; First posted 2022-05-19 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Flumazenil Adverse Reaction; Ambulatory Surgery; Postoperative Nausea; Remimazolam
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Flumazenil

STUDY DESIGN:
Intervention Model Description: Participants are administered either flumazenil (group flumazenil) or 0.9% normal saline (group control).
Who Masked: Participant, Outcomes Assessor
Masking Description: participants and outcome assessors are blinded to which group participants are allocated.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group Control (Placebo Comparator): participants are administered 2mL of 0.9% placebo at the end of procedure.
  Interventions: Drug: Flumazenil
- group Flumazenil (Active Comparator): participants are administered 0.2mg (2mL) of flumazenil at the end of procedure.
  Interventions: Drug: Flumazenil

INTERVENTIONS:
Drug: Flumazenil — During the procedure, continuous infusion of remimazolam dose of 2mg/kg/hr. when procedure ends, infusion remimazolam stops and 0.9% normal saline or 0.2mg of flumazenil according to allocated groups.
  Other Names: placebo

SUMMARY:
Remimazolam, a brand-new sedative which has benzodiazepine property. It is an ultra-short acting sedative and regarded as a proper drug for procedural sedation.

DETAILED DESCRIPTION:
As ambulatory surgery has been increased last two decades, 'Enhanced Recovery After Surgery (ERAS)' also has become an important issue in clinical fields.

It is very critical that managing postoperative pain, postoperative nausea and vomiting (PONV) and rapid recovery with less complication or side effect to anesthesiologists.

Even though remimazolam considered as an ultra-short acting sedative, it shows a relatively longer recovery time than propofol. Fortunately, remimazolam has its own antidote, called 'flimazenil'. With flumazenil, the time to recovery of consciousness dramatically reduces.

Common side effects of flumazenil include headache, dizziness, nausea, vomiting, flushing, sweating and injection pain.

In this trial we would like to demonstrate that routine single dose of flumazenil could be administered as an antidote of remimazolam without complications or side effects in gynecologic ambulatory surgery.

ELIGIBILITY:
Inclusion Criteria:

* participants aged over 20 years scheduled for ambulatory gynecologic surgery.

Exclusion Criteria:

* allergy or hypersensitivity to flumazenil, benzodiazepines, NSAIDs, 5-HT3
* arrhythmia, myocardial infarction, coronary artery disease
* obstructive sleep apnea
* severe or acute respiratory distress
* tricyclic anti-depressant
* lactose intolerance
* BMI over 30kg/m2
* ASA classification 4 or 5

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2022-08-02 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-05-13 (Actual)

PRIMARY OUTCOMES:
the incidence of postoperative nausea and vomiting (PONV) | up to 24 hours after participants discharge from day surgery center.
  assess PONV with ordinal scale; 0=none, 1= nausea, 2= retching, 3=vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Seong-Hyop Kim, M.D. Ph.D, Principal Investigator — Konkuk University Medical Centre
Locations (1):
- Konkuk University Medical Center, Seoul, Seoul-T'ǔkpyǒlshi, South Korea

IPD SHARING:
Plan to Share IPD: No